CLINICAL TRIAL: NCT00775502
Title: Open-Label, Multi-Center, Dose Escalation Phase 1/2 Study of Anti-GM2 Ganglioside Monoclonal Antibody BIW-8962 as Monotherapy in Subjects With Previously Treated Multiple Myeloma
Brief Title: Phase 1/2 Study of Anti GM-2 Monoclonal Antibody To Treat Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of efficacy in Multiple myeloma
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIW-8962-001
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; GM-2 ganglioside; monoclonal antibody; Potelligent design; Treatment of subjects who have failed previous treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — BIW-8962

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIW-8962, monoclonal antibody (Experimental)
  Interventions: Drug: BIW-8962

INTERVENTIONS:
Drug: BIW-8962 — Intravenous administration of liquid dosage form. Doses 0.03, 0.10, 0.30, 1.0, 3.0, and 10 mg/kg. Frequency is once every two weeks. Duration is 6 months
  Other Names: anti GM2 monoclonal antibody

SUMMARY:
This study will test the ability of a specially designed monoclonal antibody to destroy multiple myeloma cells. This antibody is unique in its ability to promote the death of multiple myeloma cells by processes known as antibody dependent cellular cytotoxicity (ADCC)and complement dependent cytotoxicity (CDC). The study is designed to determine both the optimal dose of the antibody to destroy multiple myeloma cells and frequency of dosing.

DETAILED DESCRIPTION:
BIW-8962 is a monoclonal antibody which targets the GM-2 ganglioside which is expressed at high levels on the surface of multiple myeloma cells. This is a Phase 1/2 study design. The Phase 1 component will establish the active biologic dose (ABD) or the maximum tolerated dose (MTD) as well as the appropriate dosing frequency based on the pharmacokinetics of the antibody and approximately 45 subjects will be enrolled in this part of the study. The initial dosing frequency will be every two weeks and the doses to be tested will range from 0.03 mg/kg to 10 mg/kg. Once the recommended Phase 2 dose and frequency have been established in Phase 1, the efficacy of the drug will be investigated in approximately 35 subjects in Phase 2.

The study did not proceed beyond the Phase 1a portion.

On 30 Nov 2010, Kyowa Hakko Kirin Pharma, Inc. (KKP) notified Investigators of the decision to terminate BIW-8962-001 due to a lack of efficacy in Multiple Myeloma.

The Phase 1 Part B and the Phase 2 components of the study were not conducted. The study was terminated and summarized in an abbreviated clinical study report (submitted 26 June 2012; SN045). Kyowa Kirin Pharma has no current plans to pursue the use of BIW8962 in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory myeloma
* M-protein in serum and/or urine by IMWG criteria.
* Bone marrow plasma cells or plasmacytoma
* Related organ or tissue impairment (CRAB)
* Subjects without detectable M protein are eligible if they have an abnormal serum free light chain ratio (FLC) or if they have at least 10% plasma cells in the bone marrow

Exclusion Criteria:

* Ongoing infection
* Cardiac disease
* Uncontrolled hypertension
* Active liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Serum M protein levels | one month

SECONDARY OUTCOMES:
Time to progression or death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zonder, MD, Principal Investigator — Karmanos Cancer Center
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Duke Medical Center, Durham, North Carolina
  - Taussig Cancer Center- Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Baz RC, Zonder JA, Gasparetto C, Reu FJ, Strout V. Phase I Study of Anti-GM2 Ganglioside Monoclonal Antibody BIW-8962 as Monotherapy in Patients with Previously Treated Multiple Myeloma. Oncol Ther. 2016;4(2):287-301. doi: 10.1007/s40487-016-0034-y. Epub 2016 Nov 2. PMID 28261656